CLINICAL TRIAL: NCT01165606
Title: Effects of Respiratory Physiotherapy in Critically Ill Patients Ventilated for More Than 48 Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Other Study IDs: Physiotherapy
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physiotherpy (Experimental)
  Interventions: Procedure: Chest physiotherapy

INTERVENTIONS:
Procedure: Chest physiotherapy

SUMMARY:
This study aimed to determine the impact of providing chest physiotherapy on the duration of mechanical ventilation, intensive care length of stay, intensive care and hospital mortality in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years, admitted to the ICU needing mechanical ventilation for longer than 48 hours

Exclusion Criteria:

* Patients with ventilatory failure due to neuromuscular dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
intensive care mortality
120-day mortality

SECONDARY OUTCOMES:
duration of mechanical ventilation
intensive care length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São José, Criciúma, Santa Catarina, Brazil